CLINICAL TRIAL: NCT01443728
Title: Vitamin D for Sickle-cell Respiratory Complications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gary M Brittenham, MD (Other)
Responsible Party: Sponsor-Investigator, Gary M Brittenham, MD, James A. Wolff Professor of Pediatrics, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAE3244; R01FD003894 (FDA)
Record Dates: First submitted 2011-09-27; First posted 2011-09-30 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Sickle Cell Disease; Vitamin D Deficiency; Acute Chest Syndrome; Asthma; Respiratory Infections
Keywords: sickle cell disease; acute chest syndrome; respiratory complications; vitamin D
MeSH Terms: conditions — Anemia, Sickle Cell; Vitamin D Deficiency; Acute Chest Syndrome; Asthma; Respiratory Tract Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 100,000 IU (Experimental): Oral vitamin D3, 100,000 IU [2.5 mg] given once a month
  Interventions: Drug: Experimental: Vitamin D3 100,000 IU
- Vitamin D3 12,000 IU (Active Comparator): Standard dose oral vitamin D3 12,000 IU [0.3 mg] given once a month
  Interventions: Drug: Active Comparator: Vitamin D3 12,000 IU

INTERVENTIONS:
Drug: Experimental: Vitamin D3 100,000 IU — Oral vitamin D3, 100,000 IU [2.5 mg] given once a month
  Other Names: Cholecalciferol
  Arms: Vitamin D3 100,000 IU
Drug: Active Comparator: Vitamin D3 12,000 IU — Standard dose oral vitamin D3 12,000 IU [0.3 mg] given once a month
  Other Names: Cholecalciferol
  Arms: Vitamin D3 12,000 IU

SUMMARY:
This study aims to answer the question whether oral vitamin D supplementation can decrease lung complications in children and adolescents with sickle cell disease. Lung complications are the leading causes of morbidity and of death in sickle cell disease. Infections and increased inflammation play important roles in the development of the lung problems in sickle cell disease. Emerging evidence shows that vitamin D helps the immune system to fight infection and to control inflammation and could potentially help prevent respiratory complications in patients with sickle cell disease. The investigators hypothesize that oral vitamin D3, 100,000 IU (2.5 mg), given once a month to a group of children and adolescents with sickle cell disease, will reduce the rate of respiratory events (infection, asthma exacerbation and acute chest syndrome) compared to the rate in a group given standard dose oral vitamin D3, 12,000 IU (0.3 mg) given once a month.

Funding Source - U.S. Food & Drug Administration, Office of Orphan Products Development

DETAILED DESCRIPTION:
This study will be a Phase 2 double-blind randomized clinical trial in 80 patients with sickle cell disease, ages 3 to 20 years-old, comparing a 2-year monthly oral dose of vitamin D3, 100,000 IU (equivalent to 3,300 IU/day) to a standard monthly dose, 12,000 IU (400 IU/day) in reducing the rate of respiratory events (defined as respiratory infections, acute asthma exacerbation, and the acute chest syndrome) in children and adolescents with sickle cell disease in comparison with the rates of respiratory events over a baseline period of one year.

Eligible participants (130 patients) will initially be screened to determine their blood vitamin D levels (serum 25-hydroxyvitamin D). Those with 25-hydroxyvitamin D levels between 5 and 60 ng/mL will be eligible for randomization. At study entry, blood and urine samples will be collected for routine and special blood tests including tests on immune function, inflammation, and bone function. Children above 5 years old will also have lung function and muscle strength tests. Participants will be followed once a month to administer the study medication (oral vitamin D3) and to monitor any side effects from the study medication by history, examination and blood and urine tests. After 12 and 24 months of therapy, the same study procedures at study entry will be repeated.

This study could help establish oral vitamin D3 as a simple, low cost treatment to reduce respiratory complications in children and adolescents with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell disease (HbSS, HbSC, HbS Beta-thalassemia)
* Age 3 to 20 years old

Exclusion Criteria:

* Patient (or parent or guardian) unwilling or unable to provide written informed consent (and assent, if applicable)
* Patient unable or unwilling to comply with requirements of the clinical trial
* Participation in other therapeutic clinical trial
* Current diagnosis of rickets
* History of hypercalcemia or diagnosis of any medical condition associated with hypercalcemia, including primary hyperparathyroidism, malignancy, sarcoidosis, tuberculosis, granulomatous disease, familial hypocalciuric hypercalcemia
* Current use of corticosteroids, excluding inhaled steroids
* Current use of anticonvulsants (phenytoin, phenobarbital, carbamazepine)
* Therapy with thiazide diuretics or lithium carbonate
* Known liver or renal disease
* Patients taking medications for pulmonary complications of sickle cell disease not on a stable dose of medications, as defined by a change in medications or doses within the three months prior to study entry
* Patients on chronic red blood cell transfusion therapy
* Absence of baseline record of respiratory events (respiratory infections, asthma exacerbations, episodes of acute chest syndrome) for the preceding year
* Pregnancy

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2011-12-13 (Actual); Primary Completion 2013-06-20 (Actual); Study Completion 2015-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Brittenham, MD, Principal Investigator — Columbia University; Margaret T. Lee, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Lee MT, Kattan M, Fennoy I, Arpadi SM, Miller RL, Cremers S, McMahon DJ, Nieves JW, Brittenham GM. Randomized phase 2 trial of monthly vitamin D to prevent respiratory complications in children with sickle cell disease. Blood Adv. 2018 May 8;2(9):969-978. doi: 10.1182/bloodadvances.2017013979. PMID 29712666

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were consented and then randomized. Only individuals who were randomized were included in the data analysis, so demographics are only available for the 62 randomized.
Pre-assignment Details: Only participants who were randomized (62) were included in the analysis of data.
Period: Overall Study
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Started | 31 | 31
Completed | 28 | 28
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (4.0) | 9.9 (3.8) | 9.9 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 15 | 15 | 30
Sickle-cell Type [Count of Participants; unit: Participants]
  SS | 26 | 28 | 54
  SC | 3 | 2 | 5
  Sb0 thalassemia | 1 | 1 | 2
  Sb1 thalassemia | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Annual Rate of Respiratory Events
Description: Defined as respiratory infection, acute asthma exacerbation, and acute chest syndrome.
Time Frame: Up to 2 years
Measure: Mean (Standard Deviation); unit: events per year
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 31 | 31
events per year
  Baseline | 3.91 (0.35) | 4.34 (0.35)
  Year 1 | 3.34 (0.37) | 4.28 (0.36)
  Year 2 | 1.54 (0.37) | 1.49 (0.37)

2. Secondary Outcome: Mean 25-Hydroxyvitamin D (25-OHD)
Description: The overall mean serum 25-OHD concentration will be measured for both groups.
Time Frame: 2 years
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 31 | 31
ng/mL | 36.1 [14 to 38] | 19.1 [13 to 20]

3. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Percent predicted forced vital capacity will be calculated for both groups.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: Percentage of predicted FVC
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 28 | 30
Percentage of predicted FVC
  Baseline | 85.5 (2.8) | 90.2 (2.3)
  Year 1 | 85.2 (2.7) | 92.4 (2.3)
  Year 2 | 85.0 (2.5) | 92.1 (2.5)

4. Secondary Outcome: Forced Expiratory Volume (FEV) in 1 Second (FEV1)
Description: Percent predicted forced expiratory volume in 1 second will be calculated for both groups.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: Percentage of predicted FEV1
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 28 | 30
Percentage of predicted FEV1
  Baseline | 80.4 (2.4) | 84.9 (2.3)
  Year 1 | 79.1 (2.7) | 85.3 (2.1)
  Year 2 | 78.9 (2.8) | 84.5 (2.0)

5. Secondary Outcome: FEV1/FVC Ratio
Description: The ratio of FEV1 to FVC will be calculated (in percentage).
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 28 | 30
ratio
  Baseline | 84.0 (1.5) | 83.3 (1.5)
  Year 1 | 82.6 (1.0) | 81.7 (1.3)
  Year 2 | 82.2 (1.5) | 81.6 (1.2)

6. Secondary Outcome: FEF 25-75
Description: Percent predicted forced expiratory flow (FEF) during expiration of 25 to 75% of the FVC will be calculated.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: Percentage of predicted FEF
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 28 | 30
Percentage of predicted FEF
  Baseline | 69.8 (5.2) | 68.8 (4.9)
  Year 1 | 62.9 (4.4) | 64.8 (4.3)
  Year 2 | 62.8 (4.4) | 65.6 (4.3)

7. Secondary Outcome: RV/TLC Ratio
Description: The ratio of residual volume (RV) to total lung capacity (TLC) will be calculated (in percentage).
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: Percent ratio
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 23 | 20
Percent ratio
  Baseline | 26.9 (1.3) | 25.1 (1.6)
  Year 1 | 25.4 (1.8) | 22.6 (1.9)
  Year 2 | 22.8 (1.6) | 21.8 (1.9)

8. Secondary Outcome: DLCO
Description: Percent predicted of the diffusing capacity for carbon monoxide in the lungs (DLCO) will be measured.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: Percentage predicted DLCO
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 20 | 19
Percentage predicted DLCO
  Baseline | 68.0 (3.2) | 72.3 (3.9)
  Year 1 | 62.9 (3.2) | 67.8 (2.4)
  Year 2 | 68.1 (3.8) | 72.9 (2.9)

9. Secondary Outcome: FeNO
Description: Fractional exhaled nitric oxide (FeNO) will be measured in parts per billion (ppb).
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 28 | 30
parts per billion
  Baseline | 19.3 (2.7) | 16.9 (2.1)
  Year 1 | 20.5 (3.5) | 16.1 (2.1)
  Year 2 | 18.1 (2.7) | 16.4 (2.4)

10. Secondary Outcome: MIP
Description: Maximum inspiratory pressure (MIP) will be measured.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: cm of water
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 23 | 19
cm of water
  Baseline | 69.1 (5.6) | 59.9 (5.3)
  Year 1 | 78.7 (6.1) | 80.4 (6.3)
  Year 2 | 77.4 (5.0) | 74.6 (4.7)

11. Secondary Outcome: MEP
Description: Maximum expiratory pressure (MEP) will be measured.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: cm of water
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 23 | 19
cm of water
  Baseline | 66.3 (3.9) | 66.3 (5.4)
  Year 1 | 60.4 (3.3) | 57.3 (3.1)
  Year 2 | 58.7 (3.4) | 56.2 (4.0)

12. Secondary Outcome: Hand-grip, Right
Description: Muscle strength was measured by looking at hand-grip strength in the right hand.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: pounds of force
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 25 | 27
pounds of force
  Baseline | 21.2 (3.2) | 16.9 (2.2)
  Year 1 | 20.6 (3.0) | 16.6 (2.4)
  Year 2 | 23.8 (4.1) | 17.4 (2.9)

13. Secondary Outcome: Hand-grip, Left
Description: Muscle strength was measured by looking at hand-grip strength in the left hand.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: pounds of force
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 25 | 27
pounds of force
  Baseline | 19.9 (3.4) | 16.0 (2.1)
  Year 1 | 19.0 (3.4) | 13.6 (2.4)
  Year 2 | 19.6 (3.6) | 15.8 (2.8)

14. Secondary Outcome: Hand-grip, Dominant
Description: Muscle strength was measured by looking at hand-grip strength in the dominant hand.
Time Frame: Up to 2 years
Population: Only includes participants who completed the assessment.
Measure: Mean (Standard Deviation); unit: pounds of force
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Number analyzed (Participants) | 25 | 27
pounds of force
  Baseline | 21.2 (3.2) | 17.1 (2.2)
  Year 1 | 20.8 (3.0) | 17.3 (2.4)
  Year 2 | 23.8 (4.1) | 18.1 (3.1)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Vitamin D3 100,000 IU | Vitamin D3 12,000 IU
Serious Adverse Events (participants affected / at risk) | 11/31 | 6/31
Other Adverse Events (participants affected / at risk) | 26/31 | 24/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D3 100,000 IU (N=31) | Vitamin D3 12,000 IU (N=31)
Acute Chest Syndrome (General disorders) | 6 | 5
Pain Syndrome (Grade 3 & 4) (General disorders) | 7 | 5
Mucosal Infection (Herpetic Gingivostomatitis) (Infections and infestations) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Cholecystitis (Gastrointestinal disorders) | 1 | 1
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecystitis (Gastrointestinal disorders) | 1 | 0
Hypoxemia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (General disorders) | 1 | 0
Sepsis (Blood and lymphatic system disorders) | 1 | 0
Varicella Zoster (Infections and infestations) | 1 | 0
Cervical Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D3 100,000 IU (N=31) | Vitamin D3 12,000 IU (N=31)
Anemia (Blood and lymphatic system disorders) | 2 | 5
Pain Syndrome (Grade 1 or 2) (General disorders) | 15 | 15
Constipation (Gastrointestinal disorders) | 2 | 0
Blood Bilirubin Increased (Blood and lymphatic system disorders) | 4 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Acute Otitis Media (Infections and infestations) | 1 | 2
Injury (Injury, poisoning and procedural complications) | 4 | 2
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Upper Respiratory Infection (Infections and infestations) | 6 | 2
Streptococcal Pharyngitis (Infections and infestations) | 2 | 5
Fever (General disorders) | 7 | 4
Acute Chest Syndrome (Grade 1 & 2) (General disorders) | 7 | 2
Influenza A/B (Infections and infestations) | 5 | 4
Acute Pharyngitis (General disorders) | 3 | 2
Seizure (General disorders) | 0 | 2
Urinary Tract Infection (Renal and urinary disorders) | 3 | 2
Headache (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes